CLINICAL TRIAL: NCT01046006
Title: Phase II Study of Combination Bortezomib, Dexamethasone, and Rituximab in Previously Untreated Patients With Waldenstrom's Macroglobulinemia: A Multicenter Trial of the European Myeloma Network
Brief Title: Bortezomib, Dexamethasone, and Rituximab in Previously Untreated Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meletios A. Dimopoulos (Other)
Collaborators: European Myeloma Network B.V. (Network)
Responsible Party: Sponsor-Investigator, Meletios A. Dimopoulos, Professor of Clinical Therapeutics, University of Athens
Organization: University of Athens (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-CAN-2021
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: lymphoma; Bortezomib; Rituximab
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma | interventions — Bortezomib; Rituximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib, Rituximab, Dexamethasone (Experimental): BDR will be administered in one 21-day treatment cycle followed by four 35-day treatment cycles to patients with WM. Bortezomib will be administered as an iv push over 3 to 5 seconds at a dose of 1.3mg/m2/day on days 1,4,8 and 11 of cycle 1. On cycles 2-5 bortezomib will be given at a dose of 1.6mg/m2/day on days 1,8,15 and 22 of each cycle. Only on cycles 2 and 5, following the administration of Bortezomib, dexamethasone 40mg iv and Rituximab 375 mg/m2 iv will be administered. A total of 8 infusions of rituximab will be administered. Subsequently patients rated as CR, PR, MR or SD will be followed without any treatment until there is evidence of progressive disease.
  Interventions: Drug: Bortezomib, Rituximab, Dexamethasone

INTERVENTIONS:
Drug: Bortezomib, Rituximab, Dexamethasone — Bortezomib as an iv push over 3 to 5 seconds at a dose of 1.3mg/m2/day on days 1,4,8 and 11 of cycle 1.
  On cycles 2-5 bortezomib will be given at a dose of 1.6mg/m2/day on days 1,8,15 and 22 of each 35-day cycle.
  Dexamethasone IV 40 mg will be given on cycles 2 and 5 on days 1,8,15,22 Rituximab IV will be given on cycles 2 and 5, 375 mg/m2, on days 1,8,15,22 iv
  Other Names: BDR

SUMMARY:
Rituximab is a monoclonal antibody with proven efficacy in WM but responses are slow. Bortezomib has shown significant and rapid activity in WM. Combinations of bortezomib with rituximab nad dexamethasone with rituximab have shown synergistic activity in laboratory studies and clinical trials. This is a Phase II multicenter study designed to evaluate the safety and efficacy of the combination of Bortezomib , Rituximab and dexamethasone (BDR). BDR will be administered in one 21-day treatment cycle followed by four 35-day treatment cycles to patients with WM. Bortezomib will be administered as an iv push over 3 to 5 seconds at a dose of 1.3mg/m2/day on days 1,4,8 and 11 of cycle 1. On cycles 2-5 bortezomib will be given at a dose of 1.6mg/m2/day on days 1,8,15 and 22 of each cycle. Only on cycles 2 and 5, following the administration of Bortezomib, dexamethasone 40mg iv and Rituximab 375 mg/m2 iv will be administered. A total of 8 infusions of rituximab will be administered. Subsequently patients rated as CR, PR, MR or SD will be followed without any treatment until there is evidence of progressive disease.

DETAILED DESCRIPTION:
Waldenstrom's macroglobulinemia (WM) is a distinct B-cell lymphoproliferative disorder characterized primarily by bone marrow infiltration with lymphoplasmacytic cells, along with demonstration of an IgM monoclonal gammopathy. This condition is considered to correspond to the lymphoplasmacytoid lymphoma as defined by the REAL2 and WHO classification systems. WM is a rare disease, with an incidence that is less frequent than multiple myeloma, and accounts for approximately 2% of all hematologic malignancies. The age-adjusted incidence rate is 3.4 per million among males and 1.7 per million among females in the US, with a geometrical increase with age. Despite continuing advances in the therapy of WM, the disease remains incurable with a median survival of 5 to 8 years from the time of diagnosis thereby necessitating the development and evaluation of novel therapeutics. Overall response rates (ORR) of 30-70% with complete response (CR) rates of up to 10% have been reported with the use of alkylator agents (e.g. chlorambucil), nucleoside analogues (cladribine or fludarabine), and the monoclonal antibody rituximab these therapeutic agents in the upfront therapy of WM with median durations of response averaging 2-3 years. Higher response rates including CR rates of up to 20% have been reported in studies combining nucleoside analogues with rituximab, and/or alkylator agents. Importantly, individual patients including the presence of cytopenias, need for more rapid disease control, age, and in particular candidacy for autologous transplant therapy should be taken into account in making the choice of first line therapy. For patients who are candidates for autologous transplant therapy, and in whom such therapy is seriously considered, exposure to alkylator or nucleoside analogue therapy should be limited. Monoclonal antibodies have been successfully used to treat patients with Waldenstrom's macroglobulinemia (WM). Most of these efforts to date have focused on the use of rituximab, a chimeric IgG1 monoclonal antibody which targets CD20, an antigen which is widely expressed in WM. Several studies employing standard dose rituximab therapy have demonstrated major response (>50% reduction in serum IgM) rates of 30%, and durations of response of about 8 months13-17. More recently, the use of extended schedule rituximab has been evaluated. Time to response after rituximab is slow and exceeds 3 months on the average. In many patients a transient increase of serum IgM may occur immediately following initiation of rituximab. Such an increase does not herald treatment failure and most patients will return to their baseline serum IgM by 12 weeks. However, patients with baseline serum IgM levels of >50g/L may be particularly at risk for a hyperviscosity-related event. Bortezomib is a small molecule proteasome inhibitor developed by Millennium Pharmaceuticals, Inc., (MPI) as a novel agent to treat human malignancies. Bortezomib is currently approved by the US FDA and by the European EMEA for the treatment of multiple myeloma. By inhibiting a single molecular target, the proteasome, bortezomib affects multiple signaling pathways. The anti-neoplastic effect of bortezomib likely involves several distinct mechanisms, including inhibition of cell growth and survival pathways, induction of apoptosis, and inhibition of expression of genes that control cellular adhesion, migration and angiogenesis. Thus, the mechanisms by which bortezomib elicits its anti-tumor activity may vary among tumor types, and the extent to which each affected pathway is critical to the inhibition of tumor growth could also differ. The mechanism of anti-tumor activity in NHL is not known; however, bortezomib inhibits the growth of various human lymphoma cell lines, as well as the survival primary WM cells. Bortezomib has been administered to patients with WM in the context of prospective studies. Chen et al administered bortezomib to 16 patients with either untreated or pretreated WM who had received ≤3 prior regimens. Six of 13 evaluable patients (46%) achieved a partial response. Dimopoulos et al administered bortezomib to 10 patients with relapsed or refractory WM. Six of these patients achieved a partial response which occurred at a median of 1 month. The median time to progression in the responding patients is expected to exceed 11months. The more common toxicities were mild or moderate thrombocytopenia, fever and fatigue; peripheral neuropathy occurred in 3 patients. The WM Clinical Trials Group (WMCTG) conducted a Phase II Study (DFCI Protocol 03-248) of single-agent bortezomib in 27 patients with relapsed or refractory WM. In an interim analysis, the safety and efficacy results for 15 patients who completed at least 2 cycles of therapy were reported.37 Eight and 7 of these patients had relapsed and refractory disease, respectively. With a median of 3 completed cycles (range 2-8), 12 of 15 (80%) patients have demonstrated a response with 5 partial responses (>50% decrease in serum IgM) and 7 minor responses (>25% decrease in serum IgM) observed. Three other patients remain with stable disease. Therapy was generally well tolerated with greater than grade II adverse events as follows: neuropathy (n=3; 20%); neutropenia (n=3; 20%); thrombocytopenia (n=1; 7%); and rash (n=1; 7%). Adverse events were generally reversible and returned to baseline after holding or dose modifying the study drug.

Bortezomib (velcade) in combination with Rituximab have been shown to act synergistically in in vitro and in vivo models. Bortezomib plus Rituximab in combination have been used in a phase 2 clinical study for previously treated patients with indolent non-Hodgkin's lymphoma. Patients received either Bortezomib 1,3mg/m2 on d1,4,8,11 q21 days (Group A), or Bortezomib 1,6mg/m2 weekly on d1,8,15,22 q35 days (Group B). Rituximab 375mg/m2 was administered weekly for 4 weeks in all patients. Response rated were similar in groups A and B, but patients in Group B (weekly bortezomib at increased dose) experienced less toxicity. Furthermore, glucocorticoids acte synergistically with Rituximab in inducing apoptosis against various malignant NHL B cell lines. A single dose of dexamethasone administered immediately before rituximab was adequate for this synergistic effect. Furthermore, we have tested this sequence in vivo in the context of a prospective trial of dexamethasone, rituximab and cyclophosphamide for previously untreated patients with WM. This combination induced responses in 74% of patients. Based on the above we investigate a combination of bortezomib, dexamethasone and rituximab (BDR) as primary treatment for patients with WM. The following points are of importance:

A) Only patients who have an indication for treatment will be included and will exclude asymptomatic patients. This is one of few multicenter trials designed specifically for WM patients who have a predefined indication for treatment.

B) By avoiding any stem cell toxic agent, we believe that we will be able to collect adequate number of blood stem cells from our patients≤70 years of age. These stem cells could be used to support high dose therapy at the time of relapse after BDR.

C) Our previous experience with single agent bortezomib indicates a median time to response of one month. Thus, by starting treatment with bortezomib alone, we believe that we will abrogate the "IgM flare" phenomenon that occurs in almost 50% of patients receiving single-agent rituximab.

D) We will limit the use of dexamethasone to one dose (40mg) just before the administration of rituximab based on in vitro data. In contrast to multiple myeloma, there is no evidence that dexamethasone is essential for the treatment of WM. Furthermore repetitive administration of dexamethasone may be associated with increased risk for opportunistic infections.

E) We plan to administer no more than 5 cycles of bortezomib in order to avoid the increased incidence of neuropathy which usually occurs with more exposure to bortezomib. Subsequently the patients will be followed with no treatment until there is evidence of progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia as defined by consensus panel one of the Second International Workshop on Waldenstrom's macroglobulinemia.1 All patients with the diagnosis of WM will be evaluable for response according to the response criteria (section 8.1)
* No prior systemic treatment for WM. Prior plasmapheresis to control hyperviscosity, is allowed. In that case baseline monoclonal protein levels for assessment of response will be the levels prior to plasmapheresis, if this is the higher value prior to treatment initiation
* Patients must have at least one of the following indications to initiate treatment as defined by "Consensus Panel Two" recommendations from the Second International Workshop on Waldenstrom's Macroglobulinemia41.

  1. Recurrent fever, night sweats, weight loss, fatigue
  2. Hyperviscosity
  3. Lymphadenopathy which is either symptomatic or bulky (≥5cm in maximum diameter)
  4. Symptomatic hepatomegaly and/or splenomegaly
  5. Symptomatic organomegaly and/or organ or tissue infiltration
  6. Peripheral neuropathy due to WM
  7. Symptomatic cryoglobulinemia
  8. Cold agglutinin anemia
  9. Immune hemolytic anemia and/or thrombocytopenia
  10. Nephropathy related to WM
  11. Amyloidosis related to WM
  12. Hemoglobin ≤10g/dL
  13. Platelet count <100x109/L
  14. Serum monoclonal protein >5g/dL even with no symptoms
* CD20 positive disease based on any previous bone marrow immunohistochemistry or flow cytometric analysis performed up to 3 months prior to enrollment.
* Karnofsky performance status >=60.
* Life-expectancy >3 months.
* Baseline platelet count >=50 10^9/L, and absolute neutrophil count >= 0.75 10^9/L.
* Meet the following pretreatment laboratory criteria at the Screening visit conducted within 28 days of study enrollment:
* AST (SGOT): >3 times the upper limit of institutional laboratory normal.
* ALT (SGPT): >3 times the upper limit of institutional laboratory normal.
* Total Bilirubin: >2 times the upper limit of institutional laboratory normal, unless clearly related to the disease.
* Calculated or measured creatinine clearance: >=30 mL/minute.
* Serum sodium >130 mmol/L.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Prior systemic treatment with WM (plasmapheresis is allowed)
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to dexamethasone, bortezomib, boron or mannitol.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Cardiac amyloidosis
* Peripheral neuropathy or neuropathic pain grade 2 or higher as defined by NCI CTCAE version 3
* Women who are pregnant. Women who are breast-feeding and do not consent to discontinue breast-feeding. Women of childbearing age who are not willing to use effective anti-conceptive methods for the duration of the study and 6 months thereafter. Men who do not consent not to father a child during the treatment period and six months thereafter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To determine the response rate [the combined complete response (CR) + partial response (PR) + minimal response (MR)] following treatment with BDR in patients with previously untreated WM. | Every cycle while on active therapy and thereafter every 3 to 4 months for up to 2 years, or until progression of disease is documented.
  Overall Response Rates

SECONDARY OUTCOMES:
determine time to progression and assess the safety and tolerability of BDR in patients with WM. | Every cycle while on active therapy and thereafter every 3 to 4 months for up to 2 years, or until progression of disease is documented.
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Meletios A Dimopoulos, MD, Principal Investigator — University of Athens, School of Medicine
Locations (4):
- Greece (2):
  - Alexandra Hospital , Department of Clinical Therapeutics, Athens, Attica
  - Laikon Hospital, Athens, Attica
- Erasmus Medical Center, Rotterdam, Netherlands
- Hospital Universitario de Salamanca, Salamanca, Spain

REFERENCES:
- See also: European Myeloma Network page for BDR in WM trial — http://www.myeloma-europe.org/index.php?bdr-wm-trial